CLINICAL TRIAL: NCT02026830
Title: The Microbiologic Profile of Diabetic Foot Infections in Turkey (TURK-DAY): Prospective Multicenter Cohort Study
Brief Title: The Microbiologic Profile of Diabetic Foot Infections in Turkey - TURK-DAY
Acronym: TURK-DAY
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Mesut MUTLUOGLU, MD, Associate Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: TURK-DAY
Record Dates: First submitted 2013-12-30; First posted 2014-01-03 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Infection
Keywords: Diabetic foot infections; microorganisms
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetic foot infection: Patients with DM (Diabetes Mellitus) presenting with a diabetic foot infection will be enrolled in the current trial to determine the causative microorganisms and their antibiotic sensitivity patterns in diabetic patients with a foot infection in Turkey.

SUMMARY:
To determine the causative microorganisms and their antibiotic sensitivity patterns in diabetic patients with a foot infection in Turkey.

DETAILED DESCRIPTION:
Recent studies have demonstrated substantial variation in the etiology of DFIs (Diabetic Foot Infections) in different regions of the world . In contrast to Western countries, studies from Asia and Africa have demonstrated that aerobic gram-negative organisms, particularly Pseudomonas aeruginosa, are far more common . The majority of current guidelines for the management of DFIs have been prepared in Western countries . Based on the results of more recent studies from the Asian continent, however, empiric antibiotic therapy for DFIs may need to be directed at organisms with substantially different antibiotic susceptibility patterns than those recommended in current guidelines. Thus, suggested antibiotic regimens for DFIs should be optimized for local clinical practice. The aim of the current trial is to provide an up-to-date view of the causative microorganisms and their antibiotic sensitivity patterns in diabetic patients with a foot infection in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Diabetes Mellitus
* Diabetic foot wound clinically diagnosed as infected

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with DM presenting with a diabetic foot infection will be enrolled in the current trial to determine the causative microorganisms and their antibiotic sensitivity patterns in diabetic patients with a foot infection in Turkey.
Sampling Method: Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Causative microorganisms and their antibiotic sensitivity patterns in diabetic patients with a foot infection in Turkey. | 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Turhan, MD, Study Director — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Locations (1):
- GATA Haydarpasa Egitim Hastanesi, Istanbul, No State Required, Turkey (Türkiye)

REFERENCES:
- [Derived] Hatipoglu M, Mutluoglu M, Turhan V, Uzun G, Lipsky BA; Turk-Day Study Group; Sevim E, Demiraslan H, Eryilmaz E, Ozuguz C, Memis A, Ay H, Arda B, Uysal S, Motor VK, Kader C, Erturk A, Coskun O, Duygu F, Guler S, Altay FA, Ogutlu A, Bolukcu S, Yildiz S, Kandemir O, Aslaner H, Polat A, Karahocagil MK, Yasar KK, Sehmen E, Kilic S, Sunbul M, Gencer S, Bozkurt F, Yanik T, Oztoprak N, Batirel A, Sozen H, Kilic I, Celik I, Ay B, Tosun S, Kadanali A, Comoglu S, Denk A, Hosoglu S, Aydin O, Elaldi N, Akalin S, Kandemir B, Akbulut A, Demirdal T, Balik R, Azak E, Sengoz G. Causative pathogens and antibiotic resistance in diabetic foot infections: A prospective multi-center study. J Diabetes Complications. 2016 Jul;30(5):910-6. doi: 10.1016/j.jdiacomp.2016.02.013. Epub 2016 Feb 21. PMID 26965794